CLINICAL TRIAL: NCT07258394
Title: A Single-Center, Randomized, Double-Blind, Placebo-Controlled Clinical Trial Evaluating the Efficacy and Safety of Dimethyl Fumarate in Preserving Islet β-Cell Function in Patients With Type 1 Diabetes Mellitus
Brief Title: Clinical Study for Dimethyl Fumarate in Preserving Islet β-Cell Function in Type 1 Diabetes Mellitus
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Nanjing Medical University (Other)
Collaborators: The First Affiliated Hospital with Nanjing Medical University (Other); Qilu Pharmaceutical (Hainan) Co., Ltd. (Industry)
Responsible Party: Principal Investigator, Yong Gu, Deputy Director of Endocrinology Dept.; Associate Chief Physician; Associate Professor; Principal Investigator, The First Affiliated Hospital with Nanjing Medical University, Nanjing Medical University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2025-SR-439
Record Dates: First submitted 2025-07-28; First posted 2025-12-02 (Actual); Last update posted 2025-12-02 (Actual); Status verified 2025-11

CONDITIONS: Type 1 Diabetes
Keywords: Type 1 Diabetes; Immunotherapy; Pancreatic Beta-Cell Function
MeSH Terms: conditions — Diabetes Mellitus, Type 1

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Dimethyl fumarate Arm (Experimental): The dosing regimen for Dimethyl fumarate enteric-coated capsules initiates at 120 mg twice daily (bid). After 7 days, the dose should be escalated to the maintenance level of 240 mg bid. This investigational product is administered concurrently with standard insulin therapy for glycemic control in Type 1 Diabetes Mellitus (T1DM).
  Interventions: Drug: Dimethyl Fumarate Enteric-coated Capsules
- Placebo Arm (Placebo Comparator): The placebo capsules initiate at a dosage of 120 mg twice daily (bid). After 7 days, the dose should be increased to the maintenance level of 240 mg bid, administered concomitantly with standard insulin-based antihyperglycemic therapy for Type 1 Diabetes Mellitus (T1DM).
  Interventions: Drug: Matching placebo capsules

INTERVENTIONS:
Drug: Dimethyl Fumarate Enteric-coated Capsules — The dosing regimen for Dimethyl fumarate enteric-coated capsules initiates at 120 mg twice daily (bid). After 7 days, the dose should be escalated to the maintenance level of 240 mg bid. This investigational product is administered concurrently with standard insulin therapy for glycemic control in Type 1 Diabetes Mellitus (T1DM).
  Arms: Dimethyl fumarate Arm
Drug: Matching placebo capsules — The placebo capsules initiate at a dosage of 120 mg twice daily (bid). After 7 days, the dose should be increased to the maintenance level of 240 mg bid, administered concomitantly with standard insulin-based antihyperglycemic therapy for Type 1 Diabetes Mellitus (T1DM).
  Arms: Placebo Arm

SUMMARY:
Purpose of the Clinical Trial:

This clinical trial aims to investigate whether dimethyl fumarate can treat adults with newly diagnosed type 1 diabetes and to evaluate the safety profile of dimethyl fumarate.

Primary Research Questions:

Does dimethyl fumarate protect pancreatic beta-cell function in adults with newly diagnosed type 1 diabetes? What medical issues may arise in individuals taking dimethyl fumarate?

Study Design:

Researchers will compare dimethyl fumarate with a placebo (an identical substance without active ingredients) to determine whether Dimethyl fumarate can effectively treat type 1 diabetes.

Participant Activities:

Take dimethyl fumarate orally twice daily for 24 weeks. Attend on-site visits every 4 weeks during the intervention period and every 12 weeks after the intervention for examinations and assessments.

Record symptoms, blood glucose control, islet function, and insulin usage throughout the trial.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects who provide written informed consent.
2. Aged 18-65 years.
3. Diagnosed with Type 1 Diabetes Mellitus (per ADA 2024 criteria).
4. Positive for ≥2 autoantibodies: Insulin autoantibody (IAA) Glutamic acid decarboxylase autoantibody (GADA) Protein tyrosine phosphatase antibody (IA-2A) Islet cell antibody (ICA) Zinc transporter 8 autoantibody (ZnT8A) Note: For IAA-positive subjects with insulin use >14 days, ≥2 additional autoantibodies must be positive.
5. Disease duration ≤100 days post-T1DM diagnosis.
6. Random C-peptide ≥ 200 pmol/L.

Exclusion Criteria:

1. Pregnancy, lactation, or women of childbearing potential not using contraception.
2. Well-controlled glycemia with oral hypoglycemic agents alone.
3. Participation in other diabetes/immune-modulating trials.
4. ALT/AST >3× upper limit of normal (ULN).
5. History of malignancy, uncontrolled autoimmune disorders, or active infections.
6. Alcohol/drug abuse, psychiatric disorders, or conditions unsuitable for trial participation.
7. Use of immunosuppressants within 12 weeks prior.
8. Participation in other drug trials within 12 weeks prior.
9. History of drug allergies, hypersensitivity, or drug addiction.
10. Any condition deemed by investigators to compromise study integrity.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2025-12-31 (Estimated); Primary Completion 2028-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Geometric mean area under the serum C-peptide curve (AUC-C-peptide), adjusted for baseline, during a 2-hour Mixed-Meal Tolerance Test (MMTT) | Intervention Week 24, and Post-intervention Weeks 24 and 52
  Participants will consume a standardized liquid meal containing fixed amounts of carbohydrate, fat, and protein. Following consumption, blood glucose, C-peptide, and glucagon levels will be measured at 0-, 30-, 60-, 90-, and 120-minute time points over a 2-hour period.

SECONDARY OUTCOMES:
Number of participants who remain C-peptide positive (peak C-peptide concentration ≥200 pmol/L after a 2-hour MMTT). | Post-intervention Week 52
  Participants will consume a standardized liquid meal containing fixed amounts of carbohydrate, fat, and protein. Following consumption, blood glucose, C-peptide, and glucagon levels will be measured at 0-, 30-, 60-, 90-, and 120-minute time points over a 2-hour period.
Changes from baseline in the geometric mean area under the C-peptide curve (AUC-C-peptide) during the 2-hour Mixed-Meal Tolerance Test (MMTT) at Intervention Week 24 and at Weeks 24 and 52 after the end of the intervention. | Intervention Week 24, and Post-intervention Weeks 24 and 52
  Participants will consume a standardized liquid meal containing fixed amounts of carbohydrate, fat, and protein. Following consumption, blood glucose, C-peptide, and glucagon levels will be measured at 0-, 30-, 60-, 90-, and 120-minute time points over a 2-hour period.
Glycemic Control Status | Intervention Week 24, and Post-intervention Weeks 24 and 52
  Hemoglobin A1c (HbA1c) levels and changes from baseline; Number of participants with poor glycemic control (HbA1c > 9%); Number of participants with good glycemic control (HbA1c < 6.5%).
Mean Daily Dose of Exogenous Insulin Used During the 7 Days Preceding Each Study Visit | Intervention Week 24, and Post-intervention Weeks 24 and 52
Incidence Rates of Hypoglycemia/Severe Hypoglycemia and Ketosis/Diabetic Ketoacidosis (DKA) | Baseline, Weeks4, 8, 12, 16, 20 and 24 During Intervention, and 12, 24, 36, and 52 Weeks After Intervention
Incidence Rates of Flushing, Abdominal Pain, Diarrhea, Nausea, Vomiting, Pruritus, Rash, Proteinuria, Erythema, and Dyspepsia | Week 4, 8, 12, 16, and 24 During Intervention
Serum Profiles of Pro-Inflammatory and Regulatory Cytokines, Along with Other Immunological Mediators | Baseline, Week 24 During Intervention, and 24,52 Weeks After Intervention
Number, Specificities, and Titers of Islet Autoantibodies | Baseline, Weeks 24 During Intervention, and 12, 24, 36, and 52 Weeks After Intervention
White Blood Cell (WBC) Subpopulation Differentiation | Baseline, Week 24 During Intervention, and 24,52 Weeks After Intervention
  including the quantity, phenotype, and functional characteristics of T cells, B cells, and natural killer (NK) cells
Incidence Rates of Elevated Aspartate Aminotransferase (AST), Elevated Total Bilirubin (TBIL), and Lymphocytopenia | Week 4, 8, 12, 16, and 24 During Intervention
Incidence Rates of Anaphylaxis, Angioedema, and Opportunistic Infections | Week 4, 8, 12, 16, and 24 During Intervention

CONTACTS AND LOCATIONS:
Locations (1):
- Deparement of Endocrinology and Metabolism, The First Affiliated Hospital with Nanjing Medical University, Nanjing, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No